CLINICAL TRIAL: NCT00180765
Title: Regulation of the Release of Inflammatory Mediators From Blood Leukocytes: A Comparison of Healthy Subjects, Healthy Smokers and Patients With COPD.
Brief Title: Regulation of the Release of Inflammatory Mediators From Blood Leukocytes
Status: Withdrawn | Type: Observational
Why Stopped: No funding for the study
Sponsor: Imperial College London (Other)
Collaborators: Asthma UK (Other)
Responsible Party: Sponsor
Other Study IDs: 01-215
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Airway Disease; Healthy Volunteers
Keywords: Leukocytes; Eosinophils; Neutrophils; Chronic Obstructive Airway Disease; Apoptosis; Signal Transduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Up to 100ml blood will be taken by venupuncture.

SUMMARY:
Chronic obstructive pulmonary disease (COPD for short) involves inflammation inside the air passages of the lungs. This inflammation might be partly responsible for the shortness of breath, cough and susceptibility to chest infections that form part of COPD. Inflammation is caused, in part, by white blood cells that are attracted from the blood into the air passages. Once inside the air passages, the white blood cells may change (or 'differentiate') and release substances that produce inflammation and attract more white cells. The hypothesis is that the lifespan of these cells may also be prolonged such that they produce more inflammatory mediators and in turn perpetuate inflammation. The cycle of inflammation may damage the lungs, so we want to see what mediators are released by white blood cells and determine if we can inhibit this effect with existing and new drugs. We would also like to see the effect of these drugs on the life-span and function of white blood cells. We will compare the behaviour and characteristics of white cells with those from healthy smokers and healthy non-smokers to find out if there is anything different about cells from COPD patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate the mechanisms that regulate the survival of blood leukocytes as well as the synthesis and release of inflammatory mediators from cells from normal individuals and subjects with COPD. The hypothesis is that in COPD the life-span of leukocytes, such as the neutrophil, is enhanced and this may contribute to inflammation, a prominent characteristic of this disease, by secreting and releasing inflammatory mediators. We also suggest that differences may exist in the sensitivity of the various leukocytes to different therapies.

Leukocytes will be purified from the peripheral venous blood of patients with COPD as well as healthy individuals. We will then investigate the effects of novel and existing therapeutic agents on leukocyte survival and inflammatory mediator synthesis and release. We will also examine the regulation and release of enzymes known to damage lung tissue. Further studies will be carried out to elucidate the signal transduction pathways that lead to the activation, altered longevity and function of leukocytes. In other experiments ribonucleic acids or RNA may be extracted form leukocytes to investigate which genes are involved. The primary objective is to identify the mechanisms that enhance leukocyte longevity and inflammatory mediator and/or enzyme synthesis and release with a view to identifying novel targets for drug therapy.

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smoking subjects: All normal volunteers will meet the following criteria:

* Age 21-70 years.
* No history of respiratory or allergic disease.
* Normal baseline spirometry as predicted for age, sex and height.
* Non-smokers.
* No history of upper respiratory tract infection in the preceding six weeks.
* Not taking regular medication

COPD subjects: COPD is diagnosed according to American Thoracic Society, European Respiratory Society and British Thoracic Society guidelines by the doctors in Professor Barnes' COPD clinic. All COPD volunteers will meet the following criteria:

* Age between 40-75 years.
* A smoking history of at least 20 pack years. ( 1 pack year = 20 cigarettes per day for 1 year)
* FEV1:FVC ratio of <0.7, post-bronchodilator FEV1 of <85% predicted, reversibility with inhaled b2-agonist of <15% of predicted FEV1: all three criteria are required.
* Current smokers or smokers who had ceased smoking for at least 6 months.
* No history of exacerbation, oral steroid or antibiotic use within the preceding 6 weeks.
* Normal serum a-1 antitrypsin level.
* No history of other respiratory or allergic disease.
* No evidence of atopy on skin prick testing to common aeroallergens (grass pollen, cat hair, house dust mite or Aspergillus fumigatus
* These tests will have already been performed as part of routine assessment in Professor Barnes' COPD clinic and we will not need to repeat them for this study.

Healthy Smokers: All healthy smoking volunteers in trials will meet the following criteria:

* Age 21-70 years.
* Smoking history of at least 10 pack years (1 pack year = 20 cigarettes per day for 1 year).
* No history of respiratory or allergic disease.
* Normal baseline spirometry as predicted for age, sex and height.
* No history of upper respiratory tract infection in the preceding six weeks.
* Not taking regular medication.

Exclusion Criteria:

Subjects will not included in this study if they meet any of the following exclusion criteria:

* Clinically significant findings in the medical history or on physical examination other than those of COPD in the COPD group.
* Pregnant women or mothers who are breastfeeding.
* Subjects who are unable to give informed consent.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-10 (Estimated); Primary Completion 2007-02 (Estimated); Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Barnes, DSc, Principal Investigator — National Heart & Lung Institute, Imperial College
Locations (1):
- National Heart & Lung Institute, Imperial College, Chelsea, London, United Kingdom